CLINICAL TRIAL: NCT05318768
Title: Association Between Physical Activity Level ，Overall Muscle Strength and Pelvic Floor Muscle Function in Women.
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Sun Xiuli, Director, Peking University People's Hospital
Other Study IDs: PKUPH7
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Pelvic Floor Disorders; Pelvic Floor Muscle Weakness
Keywords: women; physical activity; overall muscle strength; hand grip strength; pelvic floor muscle strength
MeSH Terms: conditions — Pelvic Floor Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, it is assumed that grip strength is associated with pelvic floor muscle strength. And the outcome of pelvic floor function can be predicted by referring to the status of pelvic floor muscle strength through the value of grip strength, which is labor-saving, time-saving and more convenient for evaluating pelvic floor muscle function. Moderate physical activity and increase the overall strength can activate the potential mechanism of pelvic floor muscle contraction at the same time may be a "core muscles" overall effect, that core muscles mainly includes transverse abdominal muscle, pelvic floor muscles and the muscles around the back, these muscles in the body movement to spontaneous collaboration contract pelvic floor muscles, enhancing pelvic floor muscle function, thus reducing the incidence of pelvic floor dysfunction.

DETAILED DESCRIPTION:
This study is a cross-sectional observational study, planned to enroll 942 participants from Gynecology Outpatient Clinic. Uniformly trained physicians as investigators to collect indicators from questionnaires and physical examinations.

Questionnaires may contain general information which include the patient's age, height, body weight before pregnancy and childbirth, weight gain during pregnancy, gestational age, pregnancy time, production time, high palace, delivery mode, neonatal birth weight, body length, blood sugar, blood fat, whether or not to use during pregnancy, childbirth, labor, perineal laceration, forceps midwifery, episiotomy and epidural data, pelvic floor cognition degree, physical activity levels, pelvic floor dysfunction score, pelvic floor functional impact score and sexual function score (including the prenatal and postnatal participants).

Physical examinations will be performed without the results of the questionnaire, including stress tests, pelvic floor POP-Q staging, pelvic floor muscle strength by palpation, vaginal relaxation degree, grip strength value, rectus abdominis separation, waist circumference, waist-hip ratio, etc.

Through univariate analysis of the general data of the patients, the related factors of female PFD were obtained, and the independent influencing factors of PFD were found by binary Logistic regression analysis (the dependent variable in this study was a dichotomous variable). The ROC curve was used to evaluate the predictive value of patients' overall strength level, physical activity level, body shape and other indicators on PFD outcome.

ELIGIBILITY:
Inclusion Criteria:

* Gynecological outpatient clinic patients
* In good condition and able to actively cooperate
* Agree to conduct the study.
* Age range: 18 to 80 years old

Exclusion Criteria:

* Patients who has a history of pelvic surgery or has had pelvic floor functional diseases
* Patients who do not have sex
* Pregnancy
* Patients who have serious medical diseases
* Patients with cardiac dysfunction or wear pacemakers
* Patients with neurological diseases and cognitive impairment who are difficult to cooperate with the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a cross-sectional observational study, planned to enroll 1143 participants from Gynecology Outpatient Clinic. PASS.15 software was used for sample size calculation. α- error level was set as 0.05, U0.05=1.96. For the main indicators, according to the epidemiological investigation of FEMALE PFD by our previous study, the comprehensive selection of PFD prevalence is 10%, and error δ=4%, calculated n=914, proposed to increase the loss rate by 20%. The sample size was about 1143.
Sampling Method: Probability Sample
Enrollment: 929 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength grading | through study completion，an average of one day
  The result was recorded using the modified Oxford Grading scale, ranging from 0 to 5, which 0 represents no discernible pelvic floor muscle contraction and 5 represents a strong pelvic floor muscle contraction.
Overall body strength measured by hand grip strength | through study completion，an average of one day
  Grip strength index is used to evaluate adult muscle strength in Chinese National Physical Fitness Standards. Grip strength is an important indicator to evaluate an individual's upper limb strength and can reflect the overall muscle strength level which was used to evaluate the overall strength of participants.
Physical activity levels | through study completion, an average of the past one week
  International Physical Activity Questionnaire score- short from is used to measure the overall physical activity level. Paticipants volunteered for the study and filled out questionnaires to rate their levels of physical activity over the past week which can represent the overall physical activity level.
Pelvic Floor Distress Inventory#PFDI-20#Questionnaire Score | through study completion， an average of the past 3 months
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is the short-form version of the Pelvic Floor Distress Inventory (PFDI).Since it is comprised of the UDI-6, POPDI-6, and the CRADI-8, the PFDI-20 includes 20 questions.The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100.The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
FSFI-6 Questionnaire Score | through study completion， an average of the past four weeks
  The 6-item Female Sexual Function Index (FSFI) is a short form of the original 19-item FSFI that measures sexual function in women.It comprises six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Desire and satisfaction items are rated on a 5-point Likert scale, ranging from 1 to 5, and the other items are rated on a 6-point Likert scale, ranging from 0 to 5. Total scores range from 2 to 30, with lower scores indicating worse sexual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Sun, PHD, Study Chair — Study Chair
Locations (1):
- Peking University Peoples Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
1. Date of disclosure of raw data: December 2023. Data content: original recorded data and research proposals;
  2. Ways or means of sharing IPDs, contact the researchers.
Supporting Information: Study Protocol, CSR
Time Frame: 2years
Access Criteria: contact the researchers